CLINICAL TRIAL: NCT05632224
Title: Retrospective Comparison of the Effects of Granisetron and Aprepitant in the Prevention of Postoperative Nausea and Vomiting in Laparoscopic Abdominal Surgery
Brief Title: Postoperative Nausea and Vomiting in Laparoscopic Abdominal Surgery
Acronym: PONV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Begüm Nemika Gökdemir, Medical Doctor, Baskent University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KA22/252
Record Dates: First submitted 2022-10-27; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Nausea; Vomiting
Keywords: postoperative nausea and vomiting; laparoscopic surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Aprepitant; Granisetron

STUDY DESIGN:
Intervention Model Description: group 1:patient who receive aprepitant group 2: patient who receive granisetron
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aprepitant (Active Comparator): Substance P inhibitor chemotherapeutic and also useable for prevention of postoperative nausea and vomiting
  Interventions: Drug: Aprepitant
- Granisetron (Active Comparator): 5- HT3( 5-hydroksitriptamine 3) antagonist drug for prevention of postoperative nausea and vomiting
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Aprepitant — The drug is given 1 hour before the start of the surgery
  Other Names: Emend
  Arms: Aprepitant
Drug: Granisetron — The drug is given 10 minutes before the patients's extubation
  Other Names: Sinarex
  Arms: Granisetron

SUMMARY:
The goal of this clinical trial is to compare frequency with postoperative nausea and vomiting in ASA( American Society of Anesthesiologists) I, II patients undergoing laparoscopic surgery.

The main question[s] it aims to answer are:

* Primary Outcome is the incidence of nausea and vomiting between 0-6 and 6-24 hours postoperatively and the need for additional antiemetics
* Secondary outcome is detection of additional analgesic needs and complications between 0-6 and 6-24 hours postoperatively.

Participants will receive aprepitant or granisetron for prevention of postoperative nausea and vomiting.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiveness of drugs used for postoperative nausea and vomiting in laparoscopic surgeries.

In the research; During the operation, the patient's vitals will be recorded intraoperative forms. Vitals are; heart rate, blood pressure, oxygen saturation, end tidal carbon dioxide levels; according to the pain level after awakening from the patient follow-up forms in the service.

The doses and times of analgesics will be screened, the frequencies of postoperative nausea, retching, vomiting, and additional antiemetic doses will be screened, respiratory depression, complications of anesthesia, arrhythmia, laryngospasm, hypo-hypertension, headache, dizziness, allergic reactions anxiety symptoms will be screened too.

we will try to emphasize which antiemetic is more effective than the other and which one has few side effects

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II patients patients undergoing laparoscopic surgery

Exclusion Criteria:

* ASA III and above patients who refused to participate in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-24 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
incidence of nausea | postoperative 24 hours
  the incidence of nausea between 0-6 and 6-24 hours postoperatively
the need for additional antiemetics | postoperative 24 hours
  the need for additional antiemetics between 0-6 and 6-24 hours postoperatively
incidence of vomiting | postoperative 24 hours
  the incidence of vomiting between 0-6 and 6-24 hours postoperatively

SECONDARY OUTCOMES:
additional analgesic need | postoperative 24 hours
  Detection of additional analgesic needs between 0-6 and 6-24 hours postoperatively.
detection of complications | postoperative 24 hours
  detection of complications between 0-6 and 6-24 hours postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No